CLINICAL TRIAL: NCT02461082
Title: Expiratory Muscle Strength Training (EMST) and Transcranial Magnetic Stimulation (TMS) for Treatment of Swallowing Disorders in Parkinson's Disease
Brief Title: EMST and TMS for Treatment of Dysphagia in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: Deutsche Parkinson Vereinigung (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PD-EMST-TMS
Record Dates: First submitted 2015-05-27; First posted 2015-06-03 (Estimated); Last update posted 2018-09-24 (Actual); Status verified 2017-10

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- EMST and sham-TMS (Other): Active expiratory muscle strength training in combination with sham transcranial magnetic stimulation
  Interventions: Device: Expiratory muscle strength training (EMST); Other: Transcranial magnetic stimulation (TMS)
- sham-EMST and TMS (Other): Sham expiratory muscle strength training in combination with active transcranial magnetic stimulation
  Interventions: Device: Expiratory muscle strength training (EMST); Other: Transcranial magnetic stimulation (TMS)
- EMST and TMS (Other): Active expiratory muscle strength training in combination with active transcranial magnetic stimulation
  Interventions: Device: Expiratory muscle strength training (EMST); Other: Transcranial magnetic stimulation (TMS)
- sham-EMST and sham-TMS (Other): Sham expiratory muscle strength training in combination with sham transcranial magnetic stimulation
  Interventions: Device: Expiratory muscle strength training (EMST); Other: Transcranial magnetic stimulation (TMS)

INTERVENTIONS:
Device: Expiratory muscle strength training (EMST) — The EMST is performed 4 weeks, 5 days per week, for 20 minutes per day, using a calibrated or sham, handheld device (EMST 150, Aspire Products, Gainesville, FL).
Other: Transcranial magnetic stimulation (TMS) — A sham or active transcranial magnetic stimulation is performed at the last 5 days of EMST training.

SUMMARY:
The purpose of the study is to examine the effectiveness of different methods for the treatment of dysphagia in Parkinson's disease (PD). More than 80% of patients suffering from PD develop dysphagia during the course of their disease leading to malnutrition, loss of life quality, weight loss and pneumonia, which is the leading cause of death in these patients. So far, only a few specific treatment approaches have been investigated in PD patients with swallowing disorders. The investigator want to compare a 4-week expiratory muscle strength training (EMST), transcranial magnetic stimulation (TMS), and combination of both with a sham therapy. Dysphagia severity before and after intervention is measured by flexible endoscopic evaluation of swallowing (FEES). For the evaluation of changes in cortical swallowing processing the investigators apply magnetoencephalography (MEG).

ELIGIBILITY:
Inclusion Criteria:

* Hoehn & Yahr stages II-IV
* Parkinson-related dysphagia
* Oral nutrition
* Ambulant setting
* No change of medication for at least 4 weeks before study inclusion

Exclusion Criteria:

* Other causes for dysphagia
* Other neurological disease potentially causing dysphagia
* Dementia (MMSE<25; Montreal cognitive assessment (MoCA)<26)
* Severe depression (BDI>19)
* Percutaneous endoscopic gastrostomy (PEG)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-05; Primary Completion 2018-04-06 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
Dysphagia severity as measured by FEES | Four weeks

SECONDARY OUTCOMES:
Cortical reorganization of swallowing process as detected by MEG | Four weeks and three month
Changes in quality of life as measured by the swallowing quality of life questionnaire (Swal-Qol) | Four weeks and three months
Dysphagia severity as measured by FEES | Three month

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Warnecke, MD, Principal Investigator — Universität Münster
Locations (1):
- Department of neurology, University Hospital of Muenster, Münster, North Rhine-Westphalia, Germany